CLINICAL TRIAL: NCT04335591
Title: A Double-blind Randomized Extension Study to Assess the Long-term Efficacy and Safety of Linzagolix in Subjects With Endometriosis-associated Pain
Brief Title: Extension to Study on Efficacy and Safety of Linzagolix for the Treatment of Endometriosis-associated Pain (EDELWEISS 6)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19-OBE2109-006
Record Dates: First submitted 2020-04-03; First posted 2020-04-06 (Actual); Results first posted 2024-04-30 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-03

CONDITIONS: Endometriosis
Keywords: Dysmenorrhea; Dyspareunia; Dyschezia; Non-menstrual pelvic pain
MeSH Terms: conditions — Endometriosis; Dysmenorrhea; Dyspareunia; Constipation | interventions — linzagolix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Linzagolix 75 mg (Experimental)
  Interventions: Drug: 75 mg linzagolix tablet; Drug: Placebo tablet to match 200 mg linzagolix tablet; Drug: Placebo capsule to match Add-back capsule
- Linzagolix 200 mg + Add-back (E2 1 mg / NETA 0.5 mg) (Experimental)
  Interventions: Drug: 200 mg linzagolix tablet; Drug: Placebo tablet to match 75 mg linzagolix tablet; Drug: Add-back capsule (E2 1 mg / NETA 0.5 mg)

INTERVENTIONS:
Drug: 75 mg linzagolix tablet — For oral administration once daily
  Arms: Linzagolix 75 mg
Drug: 200 mg linzagolix tablet — For oral administration once daily
  Arms: Linzagolix 200 mg + Add-back (E2 1 mg / NETA 0.5 mg)
Drug: Placebo tablet to match 75 mg linzagolix tablet — For oral administration once daily
  Arms: Linzagolix 200 mg + Add-back (E2 1 mg / NETA 0.5 mg)
Drug: Placebo tablet to match 200 mg linzagolix tablet — For oral administration once daily
  Arms: Linzagolix 75 mg
Drug: Add-back capsule (E2 1 mg / NETA 0.5 mg) — For oral administration once daily
  Arms: Linzagolix 200 mg + Add-back (E2 1 mg / NETA 0.5 mg)
Drug: Placebo capsule to match Add-back capsule — For oral administration once daily
  Arms: Linzagolix 75 mg

SUMMARY:
The primary objective of this extension study is to assess the maintenance of efficacy of linzagolix administered orally once daily for up to an additional 6 months (for up to 12 months of treatment in total) in women who have already completed 6 months of linzagolix treatment at a dose of 75 mg alone or of 200 mg in combination with ABT (E2 1 mg / NETA 0.5 mg), in the management of moderate to severe endometriosis-associated pain (EAP) in women with surgically confirmed endometriosis.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind study. Subjects who have completed the 6-month Treatment Period in 18-OBE2109-003 - Edelweiss 3 study (herein referred to as main study) will be invited to enter the present extension study. Month 6 visit of the main study is a decision point for Subjects to either end treatment and enter a post-treatment follow up (part of the main study), or to opt for a 6-month treatment extension.

All subjects will receive once daily either linzagolix 75 mg alone (with ABT placebo) or 200 mg combined with ABT for 6 months. Subjects who received placebo during the main study will be randomized to either linzagolix 75 mg alone (with ABT placebo) or linzagolix 200 mg with ABT. Subjects who received active treatment during the main study will continue with the same treatment. Double-dummy design will be used in order to maintain the blinding of the study.

After end of treatment in the extension study (6-month treatment period: from Month 6 to Month 12), subjects will enter a post-treatment Follow-Up Period of 6 months with no investigational medicinal product (IMP) or - for subjects willing to continue treatment - a second extension study will be proposed.

ELIGIBILITY:
Inclusion Criteria:

The subject must have:

* completed the 6-month treatment in the main study.
* agree to continue to use only the analgesic rescue medication permitted by the protocol during the Treatment and Follow-up Periods.
* To continue to comply with the requirements of the study protocol for the duration of the extension study.

Exclusion Criteria:

The subject will be excluded if she:

* Is pregnant or breast feeding or is planning a pregnancy within the duration of the of the study (including the Follow-up Period).
* likely to require treatment during the study with any of the restricted medications
* has any other clinically significant gynecologic condition identified during the main study on transvaginal ultrasound (TVUS), on endometrial biopsy or at the manual breast examination, which might interfere with the study efficacy and safety objectives.
* met any of the main study discontinuation criteria

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females Only
Enrollment: 356 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lecomte, Study Director — ObsEva SA
Locations (47):
- United States (8):
  - Choice Research, LLC/ ID # 609, Dothan, Alabama
  - Universal Axon - Homestead, LLC/ ID # 620, Homestead, Florida
  - Stedman Clinical Trials/ ID # 612, Tampa, Florida
  - Advanced Specialty Research/ ID # 610, Nampa, Idaho
  - Women's & Family Care, LLC dba GTC Research/ ID # 608, Shawnee Mission, Kansas
  - Southern Clinical Research / ID # 611, Metairie, Louisiana
  - Chattanooga Medical Research LLC/ ID# 602, Chattanooga, Tennessee
  - Tanner Clinic/ ID # 624, Layton, Utah
- Salzburger Landeskliniken / ID # 105, Salzburg, Austria
- Bulgaria (5):
  - Multiprofile Hospital for Active Treatment Sliven/ ID # 131, Sliven
  - MHAT Dr. Bratan Shukerov / ID #138, Smolyan
  - Medical Centre Excelsior /ID # 135, Sofia
  - Group Practice for Specialized Medical Assistance in GINART/ ID # 132, Sofia
  - University Multiprofile Hospital for Active Treatment "Sofiamed"/ ID # 133, Sofia
- Czechia (2):
  - Gynekologicko - Porodnicka Ambulance/ ID # 162, Tábor
  - Gynekologie MU Dr.Lubomir Mikulasek / ID # 160, Újezd nad Lesy
- Clinique Pasteur / ID # 206, Toulouse, France
- Poland (11):
  - Lubelskie Centrum Diagnostyczne/ ID # 402, Świdnik, Lublin Voivodeship
  - Prywatna Klinika Ginekologiczno - Położnicza/ ID # 404, Bialystok, Podlaskie Voivodeship
  - Indywidualna Specjalistyczna Praktyka Lekarska Krzysztof Wilk/ ID # 411, Katowice
  - Clinical Medical Research sp. Z o. O/ ID # 406, Katowice
  - Niepubliczny Zaklad Opieki Zrowotnej GynCentrum/ ID # 407, Katowice
  - Kotarski Jan Specjalistyczny Gabinet Ginekologiczno Polozniczy/ ID # 405, Lublin
  - Centrum Medyczne Chodźki Lublin/ ID # 403, Lublin
  - VITA LONGA Sp. z o.o./ ID # 408, Lublin
  - Centrum Ginekologii Endokrynologii i Medycyny Rozrodu "Artemida"/ ID # 409, Olsztyn
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu/ ID # 410, Przemyśl
  - Specjalistyczny Gabinet Lekarski Krzysztof Dynowski / ID # 401, Warsaw
- Romania (6):
  - Quantum Medical Center SRL/ ID # 353, Bucharest
  - Centrul Medical EUROMED/ ID # 351, Bucharest
  - Spitalul Clinic "Nicolae Malaxa"/ ID # 352, Bucharest
  - Sp Cl de Obstetrica si Ginecologie "Prof. Dr. Panait Sirbu"/ ID # 354, Bucharest
  - Gine Plus SRL Cluj- Napoca/ ID # 357, Cluj-Napoca
  - Centrul Medical GALENUS/ ID # 355, Târgu Mureş
- Spain (2):
  - Hospital Regional Universitario de Málaga/ ID # 303, Málaga
  - Hospital General Universitario Reina Sofia/ ID # 304, Murcia
- Ukraine (11):
  - City clinical maternity hospital №1/ ID # 502, Chernivtsi
  - Ivano-Frankivsk regional perinatal center, Family planning center/ ID # 506, Ivano-Frankivsk
  - Kyiv City Maternity Hospital #6/ ID # 504, Kyiv
  - Medical center of LLC "Medical Center "Verum"/ ID # 503, Kyiv
  - Institute of Pediatrics Obstetrics and Gynecology/ ID # 508, Kyiv
  - Kyiv City Clinical Hospital #9/ ID # 501, Kyiv
  - Kyiv City Center of Reproductive and Perinatal Medicine/ ID # 509, Kyiv
  - Ternopil' Communal City Hospital#2 / ID # 511, Ternopil
  - Vinnytsia City Clinical Hospital "Center of Mother and the Child "/ ID # 510, Vinnytsia
  - Zaporizhzhya Regional Clinical Hospital/ ID # 505, Zaporizhzhya
  - Maternity Hospital № 3/ ID # 507, Zaporizhzhya

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 356 subjects entered the extension study and were treated. With the exception of 3 subjects who met a discontinuation criterion at Month 6, all other subjects who entered the extension study were included in the TEAS. The PP EAS consisted of 336 subjects. All 356 subjects who entered the extension study were included in the ESAF.
Pre-assignment Details: Subjects who received placebo in the main study were randomized in a 1:1 ratio to either linzagolix (=LGX) 75 mg alone (with Add-back (=ABT) placebo) or LGX 200 mg with ABT, as per the main study randomization schedule. Subjects who received active treatment continued with the same treatment (LGX 75 mg alone or LGX 200 mg with ABT).
Groups:
- LGX 75 mg: [Main study: 6 months] The IMPs mentioned below were administered once daily orally.
  * 1 x LGX 75 mg tab.
  * 1 x LGX 200 mg placebo tab.
  * 1 x ABT placebo cap.
  [Extension study: 6 months]
  * 1 x LGX 75 mg tab.
  * 1 x LGX 200 mg placebo tab.
  * 1 x ABT placebo cap.
- LGX 200 mg+ABT: [Main study: 6 months] The IMPs mentioned below were administered once daily orally.
  * 1 x LGX 200 mg tab.
  * 1 x LGX 75 mg placebo tab.
  * 1 x ABT cap. (E2 1 mg / NETA 0.5 mg)
  [Extension study: 6 months]
  * 1 x LGX 200 mg tab.
  * 1 x LGX 75 mg placebo tab.
  * 1 x ABT cap. (E2 1 mg / NETA 0.5 mg)
- Placebo / LGX 75 mg: [Main study: 6 months] The IMPs mentioned below were administered once daily orally.
  * 1 x LGX 75 mg placebo tab.
  * 1 x LGX 200 mg placebo tab.
  * 1 x ABT placebo cap.
  [Extension study: 6months]
  * 1 x LGX 75 mg tab.
  * 1 x LGX 200 mg placebo tab.
  * 1 x ABT placebo cap.
- Placebo / LGX 200 mg+ABT: [Main study: 6 months] The IMPs mentioned below were administered once daily orally.
  * 1 x LGX 75 mg placebo tab.
  * 1 x LGX 200 mg placebo tab.
  * 1 x ABT placebo cap
  [Extension study: 6 months]
  * 1 x LGX 200 mg tab.
  * 1 x LGX 75 mg placebo tab.
  * 1 x ABT cap. (E2 1 mg / NETA 0.5 mg)
Period: Overall Study
Arm/Group | LGX 75 mg | LGX 200 mg+ABT | Placebo / LGX 75 mg | Placebo / LGX 200 mg+ABT
Started | 119 | 122 | 58 | 57
Completed | 101 | 110 | 49 | 50
Not Completed | 18 | 12 | 9 | 7
Not completed — Adverse Event | 5 | 2 | 3 | 2
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 4 | 4 | 5
Not completed — Subject planning pregnancy | 0 | 1 | 0 | 0
Not completed — Ukrainian Russian war conflict | 4 | 5 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- LGX 75 mg: [Main study: 6 months] The IMPs mentioned below were administered once daily orally.
  * 1 x Linzagolix 75 mg tab.
  * 1 x Linzagolix 200 mg placebo tab.
  * 1 x ABT placebo cap.
  [Extension study: 6 months] Same treatment as the main study
- LGX 200 mg+ABT: [Main study: 6 months] The IMPs mentioned below were administered once daily orally.
  * 1 x Linzagolix 200 mg tab.
  * 1 x Linzagolix 75 mg placebo tab.
  * 1 x ABT cap. (E2 1 mg / NETA 0.5 mg)
  [Extension study: 6 months] Same treatment as the main study
- Placebo/LGX 75 mg: [Main study: 6 months] The IMPs mentioned below were administered once daily orally.
  * 1 x Linzagolix 75 mg placebo tab.
  * 1 x Linzagolix 200 mg placebo tab.
  * 1 x ABT placebo cap.
  [Extension study: 6months] Same treatment as LGX 75 mg group in the extension study
- Placebo/LGX 200 mg+ABT: [Main study: 6 months] The IMPs mentioned below were administered once daily orally.
  * 1 x Linzagolix 75 mg placebo tab.
  * 1 x Linzagolix 200 mg placebo tab.
  * 1 x ABT placebo cap
  [Extension study: 6 months] Same treatment as LGX 200 mg+ABT group in the extension study
- Total: Total of all reporting groups
Arm/Group | LGX 75 mg | LGX 200 mg+ABT | Placebo/LGX 75 mg | Placebo/LGX 200 mg+ABT | Total
Number analyzed (Participants) | 119 | 122 | 58 | 57 | 356
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 119 | 122 | 58 | 57 | 356
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.1 (6.3) | 34.8 (6.9) | 34.3 (6.6) | 35.0 (7.7) | 34.8 (6.8)
Age, Customized [Median (Inter-Quartile Range); unit: Years] | 35.0 [31.0 to 40.0] | 35.0 [29.0 to 40.0] | 34.5 [30.0 to 40.0] | 36.0 [30.0 to 41.0] | 35.0 [30.0 to 40.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 122 | 58 | 57 | 356
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 1 | 0 | 8
  Not Hispanic or Latino | 117 | 117 | 57 | 57 | 348
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 1 | 3
  White | 117 | 120 | 58 | 56 | 351
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 0 | 0 | 1 | 0 | 1
  Romania | 6 | 7 | 4 | 3 | 20
  Czechia | 1 | 3 | 0 | 0 | 4
  Ukraine | 59 | 50 | 30 | 24 | 163
  Poland | 46 | 51 | 21 | 27 | 145
  Bulgaria | 2 | 3 | 0 | 1 | 6
  Spain | 1 | 0 | 0 | 0 | 1
  United States | 4 | 8 | 2 | 2 | 16
Weight [Mean (Standard Deviation); unit: kg] | 68.475 (15.115) | 65.210 (13.497) | 64.004 (11.103) | 68.029 (13.826) | 66.560 (13.830)
BMI [Mean (Standard Deviation); unit: kg/m2] | 24.79 (5.54) | 23.81 (4.58) | 23.39 (4.01) | 24.77 (5.06) | 24.22 (4.93)

OUTCOME MEASURES:

1. Primary Outcome: Dysmenorrhea
Description: Proportion of subjects with reduction of DYS (Month 3 MCT) and stable or decreased use of analgesics for EAP at Month 12
Time Frame: 6-month extension study treatment period (from Month 6 to Month 12)
Measure: Count of Participants; unit: Participants
Arm/Group | LGX 75 mg | LGX 200 mg+ABT | Placebo/LGX 75 mg | Placebo/LGX 200 mg+ABT
Number analyzed (Participants) | 111 | 111 | 57 | 55
Participants | 62 | 101 | 32 | 43

2. Primary Outcome: Non-menstrual Pelvic Pain
Description: Proportion of subjects with reduction of NMPP (Month 3 MCT) and stable or decreased use of analgesics for EAP at Month 12
Time Frame: 6-month extension study treatment period (from Month 6 to Month 12)
Measure: Count of Participants; unit: Participants
Arm/Group | LGX 75 mg | LGX 200 mg+ABT | Placebo/LGX 75 mg | Placebo/LGX 200 mg+ABT
Number analyzed (Participants) | 111 | 111 | 57 | 55
Participants | 66 | 75 | 34 | 27

ADVERSE EVENTS:
Time Frame: 6-month extension study treatment period (from Month 6 to Month 12)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical trial subject administered an investigational medicinal product (IMP) and which did not necessarily have a causal relationship with this treatment. Therefore, AE was any unfavorable sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an IMP, whether or not considered related to the IMP.
Arm/Group | LGX 75 mg | LGX 200 mg+ABT | Placebo/LGX 75 mg | Placebo/LGX 200 mg+ABT
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/122 | 0/58 | 0/57
Serious Adverse Events (participants affected / at risk) | 3/119 | 0/122 | 0/58 | 1/57
Other Adverse Events (participants affected / at risk) | 26/119 | 19/122 | 15/58 | 13/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LGX 75 mg (N=119) | LGX 200 mg+ABT (N=122) | Placebo/LGX 75 mg (N=58) | Placebo/LGX 200 mg+ABT (N=57)
Genital haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LGX 75 mg (N=119) | LGX 200 mg+ABT (N=122) | Placebo/LGX 75 mg (N=58) | Placebo/LGX 200 mg+ABT (N=57)
Hot flush (Vascular disorders) | 4 (4) | 5 (5) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 3 (3) | 3 (6) | 3 (4)
Anaemia (Blood and lymphatic system disorders) | 7 (7) | 0 (0) | 3 (4) | 2 (4)
Vaginal haemorrhage (Reproductive system and breast disorders) | 3 (4) | 3 (5) | 1 (1) | 3 (7)
COVID-19 (Infections and infestations) | 6 (6) | 6 (6) | 1 (1) | 2 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/91/NCT04335591/Prot_002.pdf
  • Statistical Analysis Plan (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT04335591/SAP_003.pdf